CLINICAL TRIAL: NCT05882643
Title: The Effect of the Deep Neuromuscular Block on the Refraction and the Oculocardiac Reflex During Strabismus Surgery in Pediatric Patients - a Prospective Randomized Controlled Trial
Brief Title: Deep Neuromuscular Blockade in Strabismus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Eun Jang, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-2303-079-1412
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- block group (Experimental): * Maintaining moderate to deep neuromuscular blockade during an intraoperative period (Train-of-four 0-3, post-tetanic count > 1)
  * Rocuronium (intravenous, 1.0 mg/kg)
  Interventions: Other: moderate to deep neuromuscular blockade
- control group (Active Comparator): * Maintaining shallow to minimal neuromuscular blockade during an intraoperative period (Train-of-four 4, post-tetanic count < 0.9)
  * Rocuronium (intravenous, 0.3 mg/kg)
  Interventions: Other: shallow to minimal neuromuscular blockade

INTERVENTIONS:
Other: moderate to deep neuromuscular blockade — * Maintaining moderate to deep neuromuscular blockade during an intraoperative period (Train-of-four 0-3 count, post-tetanic count > 1)
  * Rocuronium (intravenous, 1.0 mg/kg at induction period)
  Arms: block group
Other: shallow to minimal neuromuscular blockade — * Maintaining shallow to minimal neuromuscular blockade during an intraoperative period (Train-of-four 4, post-tetanic count < 0.9)
  * Rocuronium (intravenous, 0.3 mg/kg at induction period)
  Arms: control group

SUMMARY:
The purpose of this study is to determine if inducing a moderate or greater neuromuscular block (TOF count 0-3) when performing a neuromuscular block in pediatric patients aged 3 to 18 years undergoing strabismus surgery under general anesthesia can reduce the incidence of the oculocardiac reflex.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between the ages of 3 and 18 who are American Society of Anesthesiologists physical classification (ASA) I, II, or III scheduled for strabismus surgery under general anesthesia.

Exclusion Criteria:

* Patients with underlying cardiovascular disease
* Patients with preoperative electrocardiograms showing conduction disturbances
* Patients with neuromuscular disease
* Any other patient who, in the opinion of the investigator, is not a good candidate for the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 2 or greater oculocardiac reflex (induced, during strabismus surgery) | During induced oculocardiac reflex test by ophthalmologists
  > 20% reduction in heart rate induced by intentional manipulation of the extraocular rectus muscle

SECONDARY OUTCOMES:
The incidence of grade 1 oculocardiac reflex (induced, during strabismus surgery) | During induced oculocardiac reflex test by ophthalmologists
  < 20% reduction in heart rate induced by intentional manipulation of the extraocular rectus muscle
The incidence of grade 2 or greater oculocardiac reflex (during strabismus surgery) | During general anesthesia for strabismus surgery (within 2 hour)
  > 20% reduction in heart rate during strabismus surgery
The incidence of grade 1 greater oculocardiac reflex (during strabismus surgery) | During general anesthesia for strabismus surgery (usually within 2 hour)
  < 20% reduction in heart rate during strabismus surgery
Number of times Rescue IV Atropine has been used for oculocardiac reflex | During general anesthesia for strabismus surgery (within 2 hour)
  Number of times Rescue IV Atropine has been used (0.02mg/kg) for oculocardiac reflex
The incidence of hypotension | During general anesthesia for strabismus surgery (within 2 hour)
  The incidence of hypotension, defined as a drop to 20% or more of baseline mean blood pressure
Postoperative nausea/vomiting | From extubation to post-anesthesia care unit stay (within 1 hour)
  Presence of postoperative nausea/vomiting as assessed in the recovery room
Results from a refraction test before strabismus surgery | Before strabismus surgery (within 12 month)
  Results from a refraction test before strabismus surgery measured at outpatient clinic
Results from a refraction test at strabismus surgery | During general anesthesia for strabismus surgery (within 2 hour)
  Results from a refraction test during strabismus surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea